CLINICAL TRIAL: NCT04994704
Title: Comparison of Postoperative Quality of Recovery (QoR)-15 Scores According to the Use of Anesthetics (Propofol vs. Remimazolam) During Total Intravenous Anesthesia in the Spine Surgery Patients
Brief Title: Comparison of Postoperative QoR-15 Scores Between Propofol and Remimazolam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3-2021-0216
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Patients Undergoing Spine Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Experimental): Propofol based total intravenous anesthesia
  Interventions: Drug: Propfol group
- Remimazolam group (Active Comparator): Remimazolam based total intravenous anesthesia
  Interventions: Drug: Remimazolam group

INTERVENTIONS:
Drug: Propfol group — Propfol group will be started and maintained total intravenous anesthesia with propofol and remifentanil under target controlled infusion (TCI) model.
  Arms: Propofol group
Drug: Remimazolam group — Remimazolam group will be started total intravenous anesthesia with remiamazolam at 6 mg/kg/h for induction, and maintained at 0.5-1.5 mg/kg/h and remifentanil under TCI model.
  Arms: Remimazolam group

SUMMARY:
Remimazolam is a ultra-short-acting benzodiazepine, and unlike conventional benzodiazepine drugs, it is rapidly metabolized in plasma and not accumulates in the body for long periods of infusion or even with high dose administration. In addition, it has no injection pain and infusion syndrome compared with propofol. In particular, there is no study to investigate overall postoperative functional recovery via QoR-15 in patients receiving TIVA using remimazolam. Therefore, rhe purpose of the study is to compare poetoperative quality of recovery (QoR)-15 scores according to the use of anesthetics for total intravenous anesthesia in the cervical spine surgery with intraoperative neurophysiological monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who aged 20-70 years with ASA-PS 1-3,
* diagnosed of ossification of the posterior longitudinal ligament or cervical spondylotic myelopathy
* intraoperative neurophysiological monitoring.

Exclusion Criteria:

* Tolerance or hypersensitivity to benzodiazepine or propofol
* Dependence or addiction to psychotropic drugs or alcohol
* Pregnant women, subjects who lack the ability to make decisions and susceptible to voluntary participation decisions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
The difference of QoR-15 scores between two groups (propofol vs. remimazolam) | postoperative day 1
  The difference of scores in the Quality of Recovery (QoR)-15 survey.Minimum value: 0, Maximum value: 150, higher scores means better.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea